CLINICAL TRIAL: NCT02597764
Title: Use of Diaphragmatic Breathing (DB) in the Management of Bladder and Bowel Disorders in Children: A Pilot Randomized Trial
Brief Title: Diaphragmatic Breathing as an Adjunctive Therapy in the Management of Children With Bladder and Bowel Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kourosh Afshar, Study Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H14-03205
Record Dates: First submitted 2015-08-27; First posted 2015-11-05 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Bladder and Bowel Disorder, Pediatric
Keywords: Diaphragmatic breathing (DB); Bladder and bowel disorders (BBD); Autonomic nervous system (ANS); Heart rate variability (HRV); Deep breathing; Randomized controlled trial (RCT)
MeSH Terms: conditions — Intestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Urotherapy (SU) (Active Comparator): Standard Urotherapy (SU): A non-invasive therapy combining cognitive, behavioral and physical therapy. The study team will explain the problem to the children and their parents and educate them on the following: proper voiding mechanics, sitting, standing positions, how and when to void, techniques on relaxing pelvic floor muscles, and avoiding straining. An assessment of bowel habits will be done and their diet and drinking/voiding habits will be modified to maintain proper hydration with timed voiding. Voiding diaries will be provided for the assessment of the bladder and bowel habits.
  Interventions: Behavioral: Standard Urotherapy
- Standard Urotherapy (SU) + Diaphragmatic Beathing (DB) (Experimental): Standard Urotherapy (SU) with the addition of Diaphragmatic Breathing (DB):
  A non-invasive breathing technique that is performed by a marked expansion of the abdomen (contracting diaphragm) rather than chest cavity during inspiration and tightening of the stomach muscles during expiration. Participants will lie on their back on a flat surface. Head is supported with a pillow and knees are bent forward supported by another pillow. Participants will place one hand on chest and the other on the abdomen, then start inhalation by moving their abdomen out against their hand, breathing in through their nose while keeping their chest and the other hand as still as possible. During expiration, the participants will tighten their abdominal muscles by forcing them inward and breathe out through pursed lips while keeping the hand on the chest as still as possible. Participants will be asked to perform this exercise for 10 minutes 3 times daily for 3 months.
  Interventions: Behavioral: Diaphragmatic Breathing; Behavioral: Standard Urotherapy

INTERVENTIONS:
Behavioral: Diaphragmatic Breathing
  Arms: Standard Urotherapy (SU) + Diaphragmatic Beathing (DB)
Behavioral: Standard Urotherapy

SUMMARY:
Urination is a result of a complex neuro-muscular coordination which involves the action and arrangement of different parts of nervous systems as well as the muscular structure of the lower part of the urinary system. When there is an abnormal pattern in bladder and bowel habits without any known neuronal lesions, the condition is called bladder and bowel disorder (BBD). The symptoms can range from the feeling of rushing to the toilet, urinary accidents to urinating much less than expected during the day.

The standard treatment for most cases of BBD starts with Standard Urotherapy (SU) which is a beneficial basic and harmless form of treatment widely used for all children with BBD. SU involves explaining of the problem to the children and their parents by the doctors and educating them on proper voiding mechanisms, sitting, and standing positions as well as how and when to void.

The purpose of this study is to explore the possibility of testing the additive effectiveness of Diaphragmatic Breathing exercise (DB) as an alternative and harmless additional treatment to SU in children with BBD.

ELIGIBILITY:
Inclusion Criteria:

1. Children with bladder and bowel disorders (BBD) will be diagnosed by the attending pediatric urologists via a combination of thorough clinical history, physical examination, BBD Questionnaire, uroflowmetric evaluation, and voiding and stool diary.

Exclusion Criteria:

1. Known anatomic or neurological lower urinary tract abnormalities such as posterior urethral valve, urethral obstruction or stricture, ectopic ureters, congenital abnormalities of the spinal cord, or any previous surgery of the lower urinary tract.
2. Current use of medication or treatments which affects bladder or ANS function. These include anti-cholinergics, anti-psychotics, anti-depressants, and neuromodulators.
3. Any conditions or disorders that would affect the cardiovascular system or the activity of the ANS.
4. Serious pulmonary issues or diaphragmatic problems that would interfere with the practice of diaphragmatic breathing technique.
5. Psychological/behavioral abnormalities severe enough to prevent the cooperation of the child with the study coordinator or the urologist.
6. Inability to provide consent.
7. Inability to speak and/or understand in English.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2015-02; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with resolved incontinence at the end of the trial in each group (SU+DB vs. SU only). | 3 months

SECONDARY OUTCOMES:
Number of withdrawals during the treatment period. | 3 months
Number of children adhering to the diaphragmatic breathing schedule that is given to them. | 3 months
  This will be measured by the information obtained from the mobile application used during the study period.
Treatment acceptability of the proposed intervention (diaphragmatic breathing). | 3 months
  This outcome will be reported based on the participants and their parents' response to the Treatment Acceptability Questionnaires.
Change in High Frequency (HF) variation of HRV from baseline to end of treatment period for both study groups. | Baseline and 3 months
  This outcome will be measured using state-of-the-art machine for recording heart rate variability.
Change in Total Power from baseline to end of treatment period for both study groups. | Baseline and 3 months
  This outcome will be calculated from the measurements obtained from state-of-the-art machine for recording heart rate variability.
Change in heart rate from baseline to end of treatment period for both study groups. | Baseline and 3 months
Change in Pre-ejection Period (PEP) from baseline to end of treatment period for both study groups. | Baseline and 3 months
  This outcome will be measured using state-of-the-art machine for recording heart rate variability.
Change in BBD score from baseline to end of treatment period for both study groups. | Baseline and 3 months
  This outcome will be reported based on participants' response to a validated 5-point Likert scale questionnaire for diagnosing BBD.
Change in Pediatric Incontinence Questionnaire (PinQ) scores from baseline to end of treatment period for both study groups. | Baseline and 3 months
Change in average urinary flow rate (a uroflowmetry parameter) from baseline to end of treatment period for both study groups. | Baseline and 3 months
  Average urinary flow rate will be measured using top-notch equipment for measuring uroflowmetry parameters. Average urinary flow rate will be reported in mL/sec.
Change in peak urinary flow rate (a uroflowmetry parameter) from baseline to end of treatment period for both study groups. | Baseline and 3 months
  Peak urinary flow rate will be measured using top-notch equipment for measuring uroflowmetry parameters. Peak urinary flow rate will be reported in mL/sec.
Change in post-void residual volume from baseline to end of treatment period for both study groups. | Baseline and 3 months
  A hand-held ultrasound device will be used for the measurement of the post-void residual volume.

CONTACTS AND LOCATIONS:
Overall Officials: Kourosh Afshar, MD, MHSc, FAAP, Principal Investigator — University of British Columbia; Mir Sohail Fazeli, MD, PhD(c), Principal Investigator — University of British Columbia; Jean-Paul Collet, MD, PhD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's and Women's Hospital, Vancouver, British Columbia, Canada